CLINICAL TRIAL: NCT03662412
Title: Phase II Study of Sirolimus in Patients With Chemo-resistant, Recurrent or Metastatic Pancreatic Cancer
Brief Title: Study of Sirolimus in Patients With Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHZU-2018-064
Record Dates: First submitted 2018-08-20; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sirolimus treatment (Experimental): Oral solution of sirolimus, 2mg, once a day. The trial will be terminated when a serious adverse reaction occurred, or the tumor progressed rapidly twice in a row, or when the patient did not want to continue.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Oral solution of sirolimus, 2mg, once a day.
  Other Names: Rapamycin

SUMMARY:
Pancreatic cancer is a highly malignant tumor of the digestive system.In China, the annual mortality/morbidity of pancreatic cancer is as high as 0.88:1, and the morbidity and mortality are still on the rise. The 5-year survival rate of pancreatic cancer patients in the United States is only 8%, among which more than 50% of patients have distant metastasis at the time of diagnosis, and the 5-year survival rate of advanced patients with distant metastasis is as low as 3%, with extremely poor prognosis. Currently there is no standard treatment for the first - and second-line treatment resistant and postoperative recurrent patients to further prolong their survival.

mammilian target of rapamycin (mTOR) is a very important serine/threonine protein kinase involved in the regulation of energy metabolism, cell growth, angiogenesis and other cellular biological processes.Rapamycin (sirolimus) is a selective inhibitor of mTOR kinase, which can inhibit the activation and proliferation of T lymphocytes to inhibit the immune response.Currently, mTOR inhibitors are also widely used in tumor treatment. Several studies have been performed to evaluate the efficacy of sirolimus in some solid tumors, and encouraging results are obtained. However, the existing studies on mTOR inhibitors and pancreatic cancer treatment are mostly phase I trials, with little evaluation of the efficacy. Therefore, the phase II clinical trial of rapamycin in the treatment of pancreatic cancer is very necessary.

In preclinical studies, investigators found that rapamycin can effectively inhibit the angiogenesis of liver Cancer led by tumor-associated macrophages (TAM), thereby inhibiting the progression of liver Cancer.In vitro experiments on pancreatic cancer showed that rapamycin can directly inhibit the proliferation of pancreatic cancer cells.After the treatment with rapamycin in the homologous xenograft tumor model of mice, it was found that the tumor growth of mice was significantly inhibited. Further analysis suggested that rapamycin not only directly inhibits tumor proliferation, but also reverses the immune suppressive microenvironment of pancreatic cancer and promotes the T-cell-mediated anti-tumor immune response.Preclinical findings suggest that rapamycin may benefit survival in pancreatic cancer patients, which makes us very interested in the efficacy of rapamycin in patients with advanced pancreatic cancer.Therefore, investigators designed this trial to evaluate the clinical efficacy of rapamycin in patients with second-line resistance and recurrence who lacked a standard treatment regimen.

DETAILED DESCRIPTION:
1. Research purpose This clinical trial was designed to evaluate the anti-tumor effect of sirolimus in patients with advanced or postoperative recurrent pancreatic cancer with second-line standard therapy resistance.
2. Grouping and sample size calculation A single-arm study was designed. Based on clinical experience and literature, the expected median survival period of patients with advanced pancreatic cancer after second-line resistance or postoperative recurrence was about 3 months, and the median survival period of such patients was expected to be extended to 6 months after the treatment with sirolimus. The significance level of statistical test was set at 0.05 and the power of test was set as 80%, the time of enrollment was set to June 2021, and the time of follow-up was set to June 2023. The follow up loss rate was predicted as 5%, and the number of cases needed to be enrolled was calculated as 36.
3. Clinical trial procedure For the cases to be included, the patient's medical history, symptoms, signs and other conditions should be examined in advance, informed consent should be obtained and signed, and the patient's age, height, weight, medical history, symptoms, signs, pathological results, tumor node metastasis (TNM) stage and other contents should be recorded.According to the test requirements, the study was designed to be limited to 5 years, and the day of oral administration of sirolimus will be set as the first day, tumor markers will be follow up every 3 weeks.Each 3-month review includes symptoms, signs, adverse events, blood routine examination, liver and kidney function, abdominal enhanced CT, liver enhanced MRI+ diffusion, and chest high-resolution CT.

   Overall survival (OS) was taken as the primary endpoint and then recorded to the secondary endpoint. All results were recorded in the case report form, clinical efficacy and safety were evaluated, and adverse events were observed.If the patient cannot come to the hospital for reexamination, follow up will be conducted by telephone, email, etc.
4. Adverse events record and report Information on non-serious adverse events that occur during treatment should be recorded on the clinical trial report form (CRF), and all serious adverse events will be recorded in the CRF report form.Few patients in this study may have serious liver and kidney function injury, may have allergy reaction, secondary hypertension, hypercholesterolemia, serious infection and so on. In view of the above possible situations, investigators will fully evaluate the liver and kidney function before treatment, and give protective drugs for organ function; And the corresponding adjuvant drugs such as blood pressure drugs, lipid-regulating drugs to prevent sirolimus side effects;The symptoms and indicators of infection were closely monitored. Once adverse events happen, report will be sent to the general manager and the head of the hospital immediately, and also to the ethics committee of adverse events within the specified time, and make unified analysis after the study.
5. Data management and statistical analysis Data recording and auditing: The observation data will be recorded by the attending physician in the case report form, and the data records shall be timely, complete, accurate and authentic.The form will be filled out in black (or blue and black), any changes will be made by the relevant personnel, and then signed and dated. The changes will not cover the original record. If possible, copy the relevant test paper and paste it on the attached page after CRF.

   Data entry: Establish data entry program and database for statistical analysis.
6. Informed consent The subject must obtain written informed consent before performing the study procedures to inform the patient of the specific content related to the study. The specific procedures for obtaining informed consent include: the patient's disease characteristics, treatment plan and related risks shall be informed in detail by the competent doctor, and the patient or legal guardian with civil capacity shall sign the informed consent after fully knowing and understanding the relevant process and risks of this study.

ELIGIBILITY:
Inclusion Criteria:

1. patients who have failed second-line chemotherapy: patients who had previously received treatment with gemcitabine-based chemotherapy failed, and received fluorouracil based chemotherapy (such as FOLFIRINOX) and had received or not received radiotherapy and failed treatment.
2. the Eastern Cooperative Oncology Group (ECOG) score is 0-1.
3. subject's informed consent, understanding and willing to cooperate with the test program and sign relevant documents.

Exclusion Criteria:

1. patients with other malignant tumors or pancreatic cancer have unclear clinical diagnosis, or there are some retroperitoneal lesions with other unclear properties.
2. complicated with uncontrollable central nervous system metastases or neoplastic meningitis.
3. complicated with serious and uncontrollable internal diseases such as severe diabetes, severe hypertension, serious infection, congestive heart failure, ventricular fibrillation, coronary heart disease with obvious symptoms or myocardial infarction in the past 6 months.
4. patients with significant renal dysfunction (serum creatinine beyond the normal range).
5. patients with significant abnormal liver function ( serum bilirubin > 1.5 times or aspartate transaminase (AST)/aspartate transaminase (ALT) > 2.5 times of the normal upper limit, > 5 times of the normal upper limit if there is liver metastasis).
6. patients with significantly abnormal white blood cell count (WBC) (neutrophils < 1500 / mu or platelet < 100 * 10 ^ 3 L/mu L or hemoglobin < 90 g/L).
7. anesthesia, radiotherapy or systemic chemotherapy were performed within the past 2 weeks.
8. drug maintenance: immunosuppressive drugs, and treatment dose of vitamin K antagonist.
9. HIV patients.
10. others: allergic history of similar drugs, pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | Up to approximately 24 months
  The duration of time from patients begin with sirolimus treatment to the time of death or the end of the study.

SECONDARY OUTCOMES:
Response rate | Assessment performed at 6 months after the first treatment
  Remission, stable or progression

OTHER OUTCOMES:
Change of carbohydrate Antigen-199 (CA-199) level | Up to 24 months, from 1 day before the first time treatment until date of first documented progression or date of death from any cause
  Change of blood CA-199 level
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to approximately 24 months
  Adverse effect rates

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, MD Ph.D, Principal Investigator — second affiliated hospital, Zhejiang University School of Medicine
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided